CLINICAL TRIAL: NCT04510597
Title: Phase III Trial of Immunotherapy-Based Combination Therapy With or Without Cytoreductive Nephrectomy for Metastatic Renal Cell Carcinoma (PROBE Trial)
Brief Title: Comparing the Outcome of Immunotherapy-Based Drug Combination Therapy With or Without Surgery to Remove the Kidney in Metastatic Kidney Cancer, the PROBE Trial
Acronym: PROBE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1931; NCI-2020-04442 (Other: NCI)
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Continued Systemic Therapy Only (Active Comparator): Nivolumab 240 mg IV 1 q 2 weeks
  OR
  Nivolumab 480 mg IV 1 q 4 weeks
  OR
  Pembrolizumab 200 mg IV 1 q 3 weeks Axitinib 5 mg oral Daily BID
  OR
  Avelumab 10 mg/kg IV 1 q 2 weeks Axitinib 5 mg oral Daily BID
  Interventions: Procedure: Cytoreductive Nephrectomy; Drug: Active Comparator
- Arm 2: Nephrectomy and Continued Systemic Therapy (Experimental): Continued systemic therapy as above, plus:
  Radical or partial nephrectomy may be performed using laparoscopic, open, or robotic approaches. Surgery should be performed within 8 weeks of randomization.
  Interventions: Procedure: Cytoreductive Nephrectomy

INTERVENTIONS:
Procedure: Cytoreductive Nephrectomy — Radical or partial nephrectomy may be performed using laparoscopic, open, or robotic approaches. Surgery should be performed within 8 weeks of randomization
Drug: Active Comparator — Nivolumab 240 mg IV 1 q 2 weeks
  OR
  Nivolumab 480 mg IV 1 q 4 weeks
  OR
  Pembrolizumab 200 mg IV 1 q 3 weeks Axitinib 5 mg oral Daily BID
  OR
  Avelumab 10 mg/kg IV 1 q 2 weeks Axitinib 5 mg oral Daily BID
  Arms: Arm 1: Continued Systemic Therapy Only

SUMMARY:
This phase III trial compares the effect of adding surgery to a standard of care immunotherapy-based drug combination versus a standard of care immunotherapy-based drug combination alone in treating patients with kidney cancer that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as nivolumab, ipilimumab, pembrolizumab, and avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Axitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Surgery to remove the kidney, called a nephrectomy, is also considered standard of care; however, doctors who treat kidney cancer do not agree on its benefits. It is not yet known if the addition of surgery to an immunotherapy-based drug combination works better than an immunotherapy-based drug combination alone in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare overall survival in participants with newly diagnosed metastatic renal cell carcinoma who are randomized to receive immune checkpoint inhibitor-based combination treatment plus cytoreductive nephrectomy versus immune checkpoint inhibitor-based combination treatment alone.

SECONDARY OBJECTIVES:

I. To compare overall survival between arms in the subset who received their assigned protocol treatment.

II. To assess complications of nephrectomy and post-randomization drug toxicities.

III. To compare objective response rate in metastatic sites between the arms in participants with measurable metastatic disease.

IV. To assess change in diameter of primary tumor at week 12 disease assessment in participants who have received pre-randomization treatment.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE:

PRE-RANDOMIZATION TREATMENT: Treatment naive patients are assigned to 1 of 3 treatment regimens per standard of care.

REGIMEN I: Patients receive nivolumab intravenously (IV) and ipilimumab IV. Treatment repeats every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV on day 1. Cycles repeat every 2-4 weeks in the absence of disease progression or unacceptable toxicity.

REGIMEN II: Patients receive pembrolizumab IV on day 1 and axitinib orally (PO) twice daily (BID) on days 1-21. Cycles repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

REGIMEN III: Patients receive avelumab IV on day 1 and axitinib PO BID on days 1-14. Cycles repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

NOTE: Some patients may have already completed the standard of care pre-randomization treatment specified above off-trial.

RANDOMIZATION TREATMENT: Between 10-14 weeks from the start of on-trial or off-trial pre-randomization treatment, patients are randomized to 1 of 2 arms.

ARM I: Patients receive nivolumab IV, pembrolizumab IV, or avelumab IV on day 1. Patients also receive axitinib PO BID. Cycles with nivolumab repeat every 2 or 4 weeks, cycles with pembrolizumab repeat every 3 weeks, and cycles with avelumab repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Within 42 days following randomization, patients undergo radical or partial nephrectomy in addition to nivolumab, pembrolizumab, avelumab, and axitinib as in Arm I in the absence of disease progression or unacceptable toxicity. Axitinib should be stopped at least 24 hours prior to surgery.

After completion of trial treatment, patients are followed up every 3 months for the first year, every 6 months for years 2 and 3, and then annually for up to 7 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION: Participants must have a histologically proven diagnosis of clear cell or non-clear cell renal cell carcinoma. Participants with collecting duct carcinoma histology are not eligible. Participants with multifocal or bilateral tumors are eligible
* STEP 1 REGISTRATION: Participants must have primary tumor in place
* STEP 1 REGISTRATION: Participants must have the following scans performed, showing clinical evidence of measurable or non-measurable metastatic disease:

  * Computed tomography (CT) scan of the chest (can be performed without contrast if CT contrast cannot be given)
  * CT of abdomen and pelvis with contrast OR magnetic resonance imaging (MRI) of the abdomen and pelvis with or without contrast

Scans must be performed within the following timeframes:

* Treatment naive participants must have scans documenting metastatic disease completed within 90 days prior to study registration
* Previously treated participants must have scans documenting metastatic disease completed within 90 days prior to first dose of systemic treatment

  * STEP 1 REGISTRATION: Participants with symptomatic metastases may have received palliative radiotherapy or receive palliative radiotherapy after registration
  * STEP 1 REGISTRATION: Participants must have no clear contraindications to nephrectomy
  * STEP 1 REGISTRATION: Participants must be offered the opportunity to participate in specimen bank. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
  * STEP 1 REGISTRATION: Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
  * STEP 1 REGISTRATION: As part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
  * STEP 2 REGISTRATION: Participants must have at least one of the following scans performed 12 weeks (+/- 2 weeks) after starting pre-randomization treatment
* CT scan of the chest (can be performed without contrast if CT contrast cannot be given)
* CT of abdomen and pelvis with contrast OR MRI of the abdomen and pelvis with or without contrast Scans must be performed within 28 days prior to randomization. Response should be assessed by comparing with a CT or MRI of the chest, abdomen and pelvis obtained prior to starting pre-randomization treatment. Participants with complete response in all metastatic sites are not eligible to randomize to Step 2

  • STEP 2 REGISTRATION: Participants must have one of the following objective statuses after 12 weeks of pre-randomization treatment
* Stable disease
* Partial response
* The treating investigator believes the patient is deriving clinical benefit from systemic therapy AND have Zubrod performance status 0-1

  * STEP 2 REGISTRATION: Participants must plan to continue the immune-based therapy received during pre-randomization treatment
  * STEP 2 REGISTRATION: Participants must be randomized on or between the 11th and 14th week of protocol-directed pre-randomization treatment therapy
  * STEP 2 REGISTRATION: Participants must have received at least one of the minimum amounts of immunotherapy:
* 2 infusions of nivolumab + 1 infusion of ipilimumab
* 2 infusions of pembrolizumab
* 2 infusions of avelumab

  * STEP 2 REGISTRATION: Participants must have a planned surgery date within 42 days of randomization
  * STEP 2 REGISTRATION: Participants must be a surgical candidate as determined by study urologist. The urology consult should be done within 42 days prior to randomization
  * STEP 2 REGISTRATION: Participants must have a complete physical examination and medical history within 28 days prior to randomization
  * STEP 2 REGISTRATION: Participants must have a Zubrod performance status of 0-1 within 28 days prior to randomization
  * STEP 2 REGISTRATION: Total bilirubin =< institutional upper limit of normal (ULN) (within 28 days prior to randomization)
  * STEP 2 REGISTRATION: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x institutional upper limit of normal (ULN) (within 28 days prior to randomization)
  * STEP 2 REGISTRATION: Serum creatinine =< 1.5 x the institutional upper limit of normal (IULN) OR measured OR calculated creatinine clearance >= 50 mL/min using the Cockcroft-Gault Formula) (must have been drawn and processed within 28 days prior to randomization)

Exclusion Criteria:

* STEP 1 REGISTRATION: Participants must not have known active brain metastases. Participants with previously treated brain metastases are eligible if participant has no neurologic signs or symptoms suggestive of brain metastasis. Brain imaging studies are not required. If brain imaging studies are performed, they must be negative for disease
* STEP 1 REGISTRATION: Participants must not have received the following prior treatment of metastatic renal cell carcinoma:

  * Treatment naive participants must not have received any prior lines of systemic therapy for metastatic renal cell carcinoma beyond the line intended as part of protocol therapy
  * Previously treated participants must not have received any systemic therapy for metastatic renal cell carcinoma beyond the one regimen received off protocol as specified in Step 1 pre-randomization treatment
* STEP 1 REGISTRATION: Participants must not have received more than the following amounts protocol-directed pre-randomization treatment:

  * Treatment naive participants must not have received any pre-randomization treatment.
  * Previously treated participants must not be planning to receive any additional treatment prior to Step 2 randomization, and must not have received more than the following amounts of pre-randomization treatment:

    * 4 infusions of nivolumab
    * 4 infusions of ipilimumab
    * 4 infusions of pembrolizumab
    * 7 infusions of avelumab
* STEP 1 REGISTRATION: Participants must not have received immunotherapy for any cancer within the following timeframes:

  * Treatment naive participants must not have received any immunotherapy within a year of registration
  * Previously treated participants must not have received any other immunotherapy within a year of the start of off protocol specified pre-randomization treatment
* STEP 1 REGISTRATION: Participants must not have a solitary kidney and not have a transplanted kidney
* STEP 1 REGISTRATION: No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, any in situ or T1 cancer, adequately treated stage I or II cancer from which the participant is currently in complete remission, or any other cancer from which the participant has been disease free for at least two years
* STEP 1 REGISTRATION: Participants must not have been previously diagnosed with a medical condition that makes them ineligible for immune based combination therapy or nephrectomy
* STEP 2 REGISTRATION: Participants must not show progression in the primary tumor. Participants who are considered to have pseudo progression are allowed
* STEP 2 REGISTRATION: Participants must not have known active brain metastases. Participants with previously treated brain metastases are eligible if participant has no neurologic signs or symptoms suggestive of brain metastasis. Brain imaging studies are not required. If brain imaging studies are performed, they must be negative for disease
* STEP 2 REGISTRATION: No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the participant is currently in complete remission, or any other cancer from which the participant has been disease free for two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2033-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization to date of death due to any cause, assessed up to 7 years.
  Analysis will be intent-to-treat. Evidence suggesting early termination of the trial and a conclusion that the cytoreductive nephrectomy (CN) approach is superior to treatment alone would be if the null hypothesis is rejected at the one-sided 0.005 level. For the second and third interim analyses, the null and alternative hypotheses with respect to survival will be tested, with superiority tested at the one-sided 0.005 level, and futility determined to be met if the (CN versus no CN) hazard ratio is greater than or equal to 1. A proportional hazards model will be fit to estimate the hazard ratio adjusting for the stratification factors as covariates in the model. Will evaluate whether each of the stratification factors are predictive factors of cytoreductive nephrectomy by placing an interaction term corresponding to each stratification factor and treatment arm in the proportional hazards survival model.

SECONDARY OUTCOMES:
Overall survival in subset who received assigned protocol treatment | From date of randomization to date of death due to any cause, assessed up to 7 years
  Will be included in the proportional hazards regression model adjusting for stratification factors as covariates.
Progression-free survival | From date of randomization to date of first documentation of progression, or death due to any cause, assessed up to 7 years
  A proportional hazards model will be used to compare progression-free survival between arms, adjusting for the stratification factors as covariates.
Objective response | Up to 7 years
  Objective response includes all confirmed and unconfirmed partial and complete responses. Baseline will be disease assessment at randomization. Response Evaluation Criteria in Solid Tumors response rates will be evaluated, excluding the primary tumor in the kidney because that disease will be removed in half the participant's post-randomization. Comparison of response rates will be performed using logistic regression with stratification factors as covariates and an indicator for treatment arm.
Change in maximum diameter of primary tumor | From the disease assessment just prior to the start of immunotherapy to the week 12 disease assessment
  Descriptive statistics will be provided including stratified results by treatment regimen received. Potential additional analyses may include assessment of the interaction between change in primary tumor and randomized treatment arm. This will be modeled as an interaction term in the proportional hazards survival model.

CONTACTS AND LOCATIONS:
Locations (387):
- United States (387):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Keck Medicine of USC Buena Park, Buena Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Keck Medicine of USC Huntington Beach, Huntington Beach, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Mills Health Center, San Mateo, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Cedars-Sinai Cancer - Tarzana, Tarzana, California
  - City of Hope Upland, Upland, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - AdventHealth Celebration, Celebration, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Loyola Center for Health at Burr Ridge, Burr Ridge, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Loyola Medicine Homer Glen, Homer Glen, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Hematology/Oncology Clinic PLLC, Baton Rouge, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Hematology Oncology - Hayes, Clinton Township, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - University of Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Kaiser Sunnyside Medical Center, Clackamas, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - George E Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Overlake Medical Center, Bellevue, Washington
  - Valley Medical Center, Renton, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bell H, Cotta BH, Salami SS, Kim H, Vaishampayan U. "PROBE"ing the Role of Cytoreductive Nephrectomy in Advanced Renal Cancer. Kidney Cancer J. 2022 Mar 15;6(1):3-9. doi: 10.3233/kca-210010. PMID 35310961
- [Derived] Kuusk T, Abu-Ghanem Y, Mumtaz F, Powles T, Bex A. Perioperative therapy in renal cancer in the era of immune checkpoint inhibitor therapy. Curr Opin Urol. 2021 May 1;31(3):262-269. doi: 10.1097/MOU.0000000000000868. PMID 33742979